CLINICAL TRIAL: NCT06541431
Title: Analytical Validation of Stream™ Platform - Sample Collection Protocol
Brief Title: Analytical Validation of Stream™ Platform
Status: Recruiting | Type: Observational
Sponsor: FluidAI Medical (Industry)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: CLS0012
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will focus on the collection of abdominal drainage fluid from study subjects.
  Subjects that undergo gastrointestinal surgery often receive a prophylactic intra-peritoneal or pelvic drain. This drain prevents buildup of fluid in the abdominal cavity after surgery. The fluid from the drain is collected in an evacuator. The fluid may be used in laboratory, or is typically discarded. This fluid will be collected daily in this study. The fluid may contain DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sample Collection Cohort: This group will contain patients that undergo gastrointestinal surgeries, namely hepatobiliary, colorectal, trauma, and acute care procedures, and received an abdominal drain. Samples of abdominal drainage fluid will be collected daily from each patient.
  Interventions: Other: Abdominal Drainage Fluid Collection

INTERVENTIONS:
Other: Abdominal Drainage Fluid Collection — Abdominal drainage fluid will be collected daily from the subjects until they are discharged from the hospital, or their abdominal/pelvic drain is removed, as determined by the treating surgeon.

SUMMARY:
The accurate monitoring of physiological parameters in postoperative patients is essential for early detection and management of potential complications. One such critical parameter is the pH of abdominal drainage fluid, which can provide valuable insights into the patient's recovery and the presence of any postoperative infections or complications after gastrointestinal surgery. The Stream™ Platform, consisting of the Origin™ inline biosensor system and supporting materials, represents a significant advancement in this area. Origin™ is designed to be integrated inline with a standard surgical drain, enabling real-time monitoring of drainage effluent characteristics, specifically pH, which represents the acidity of the fluid.

This protocol details the analytical validation of the Stream™ Platform, focusing on the pH measurements conducted by the Origin™ device. The study aims to establish the precision, linearity, and analytical specificity of the Origin™ system. Additionally, method comparison studies will be conducted to evaluate the performance of the Origin™ device against standard bench-top comparators.

The multi-center study will be conducted using commercially available calibration fluids and abdominal drainage samples collected from patients undergoing abdominal surgeries. These samples, which include those from colorectal, hepatobiliary, and trauma and acute care patients, will be utilized to validate the Origin™ device's capability to deliver accurate and reliable pH measurements.

DETAILED DESCRIPTION:
This is a multi-center study, being conducted to facilitate the Analytical Validation of Stream™ Platform. This includes precision evaluation assessing repeatability and reproducibility of the pH measurements conducted by Origin™, tests evaluating the linearity of measurements, analytical specificity (interference testing), and method comparison studies. The tests described under this study will be completed using commercially available calibration fluids, and peritoneal drainage samples collected from patients that undergo gastrointestinal surgery. Simulated peritoneal fluids, adjusted to the required pH may be utilized in some cases. Additionally, peritoneal drainage samples may be used for testing, verification, and validation of novel Origin™features, designed to improve user workflow. The following patient populations will be eligible for the collection of abdominal drainage samples: colorectal, hepatobiliary, and trauma and acute care patients.

This study will require collection of peritoneal drainage fluid of subjects that undergo gastrointestinal surgery. One sample will be collected per day and will be labelled with a study ID, date and time of collection, and then frozen. The sample will be supplied to FluidAI team. The team at FluidAI will conduct the laboratory assessments required for analytical validation of pH measurements of Origin™.

This study does not pose any risk to participants as abdominal drainage fluid is routinely discarded as it is considered a waste product. No personal health information will be collected from the participants, and the study requires no follow up. Participation from subjects will be deemed complete when they are discharged from the hospital, or when their abdominal drain is removed as determined by their surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years - male or female
* Subject understands and has voluntarily signed and dated Informed Consent Form (ICF)
* Subjects must be willing to comply with trial requirements
* Subject has performed an open or laparoscopic surgery with abdominal/ pelvic drainage

Exclusion Criteria:

* Subject is expected to be discharged less than 8 hours post-surgery
* Subject carries has a known infectious disease such as Hepatitis B or C, HIV, TB, infections caused by multi-drug resistant organisms, or known parasitic infections affecting the gastrointestinal tract
* Involvement in the planning and conduct of the clinical investigation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects included in this study will consist of several patient populations who have undergone abdominal surgery and received an abdominal drain. This includes colorectal, hepatobiliary, and trauma and acute care patients. All subjects must meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Conduct precision evaluation of pH measurements obtained using Origin™ | 8 months
  The objective of these tests is to assess the ability of the Origin™ to provide a measurement proportional to the measurand being quantified over a defined range of pH with acceptable levels of variance, such that the device meets predefined acceptance criteria for precision estimates.
Evaluate the linearity of pH measurements obtained using Origin™ | 8 months
  The objective of this test is to establish, verify and demonstrate the linear range of Origin™ in measuring the pH of peritoneal fluid.
Evaluate the Analytical Specificity of pH measurements obtained using Origin™ | 8 months
  The objective of this test is to evaluate the effect of potential interfering substances on the clinical and analytical performance of the Origin™ via paired difference testing. In the event of an interference effect a dose-response experiment will be conducted to determine the magnitude of interference as a function of interferent concentration.
Conduct method comparison studies for measuring pH of abdominal drainage fluid | 8 months
  The objective of this test is to compare the pH measurements of abdominal drainage fluid using Origin™ and a standard benchtop comparator.

SECONDARY OUTCOMES:
Testing, verification of validation of new Origin™ features | 8 months
  To utilize samples of abdominal drainage for testing, verification and validation of new features developed to optimize the user workflow of Origin™ in hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Pablo Serrano, MD MPH FACS, Principal Investigator — Juravinski Hospital - Hamilton Health Sciences
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No